CLINICAL TRIAL: NCT03151044
Title: A Prospective, Open, Randomized Controlled, Multi-center Phase III Clinical Trial Comparing High-dose Epirubicin and Standard-dose Epirubicin in R±CEOP in Newly Diagnosed Young Patients With Medium/High-risk Diffuse Large B-cell Lymphoma
Brief Title: R±CEOP90 Versus R±CEOP75 in Newly Diagnosed Young Patients With Medium/High-risk DLBCL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: FENG Ji-feng (Other)
Collaborators: Chinese Anti-Cancer Association (Other)
Responsible Party: Sponsor-Investigator, FENG Ji-feng, Director of the hospital, Jiangsu Cancer Institute & Hospital
Organization: Jiangsu Cancer Institute & Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015NL-078
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: epirubicin; high-dose; Diffuse Large B-cell Lymphoma; medium/high-risk
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPI-90 (Experimental): Participants in this arm shall be given high-dose Epirubicin Combined with CVP ± Rituximab for six 21-day cycles:
  High-dose Epirubicin 90mg/m2, i.v., Day 1; Cyclophosphamide 750mg/m2, i.v., Day 1; Vincristine 1.4mg/m2, i.v., Day 1; Prednisolone 100mg/m2, p.o., Day 1-5;
  Plus/not plus:
  Rituximab 375mg/m2, i.v., Day 0
  Interventions: Drug: High-dose Epirubicin Combined with CVP ± Rituximab
- EPI-75 (Active Comparator): Participants in this arm shall be given standard-dose Epirubicin, Combined with CVP ± Rituximab for six 21-day cycles:
  Standard-dose Epirubicin 75mg/m2, i.v., Day 1; Cyclophosphamide 750mg/m2, i.v., Day 1; Vincristine 1.4mg/m2, i.v., Day 1; Prednisolone 100mg/m2, p.o., Day 1-5;
  Plus/not plus:
  Rituximab 375mg/m2, i.v., Day 0
  Interventions: Drug: Standard-dose Epirubicin Combined with CVP ± Rituximab

INTERVENTIONS:
Drug: High-dose Epirubicin Combined with CVP ± Rituximab — Experimental group shall be given high-dose Epirubicin (90mg/m2) combined with standard-dose Cyclophosphamide (750mg/m2), Vincristine (1.4mg/m2) and Prednisolone (100mg/m2) ± Rituximab
  Other Names: R±CEOP90
  Arms: EPI-90
Drug: Standard-dose Epirubicin Combined with CVP ± Rituximab — Active comparator group shall be given standard-dose Epirubicin and standard-dose Cyclophosphamide (750mg/m2), Vincristine (1.4mg/m2) and Prednisolone (100mg/m2) ± Rituximab
  Other Names: R±CEOP75
  Arms: EPI-75

SUMMARY:
This clinical trial is designed to compare the efficacy and safety of R±CEOP90 containing high-dose epirubicin and R±CEOP75 containing standard epirubicin in newly diagnosed young patients with medium/high-risk diffuse large B-cell lymphoma. Half of the participants receive R±CEOP regimen containing 90mg/m2 epirubicin, while the other half of participants receive R±CEOP regimen containing 75mg/m2 epirubicin. Via exploring whether high-dose epirubicin shall achieve better efficacy and less toxicity, we hope to optimize current treatment choice for young patients with medium/high-risk diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
STUDY BACKGROUND Anthracyclines are key drugs in combined chemotherapy regimen for the treatment of diffuse large B-cell lymphoma (DLBCL) and R±CHOP has been used as the first-line standard chemotherapy protocol of DLBCL. Epirubicin (EPI) belongs to anthracyclines and its mechanism of action includes directly embedding into DNA base pair, interfering with the transcription process, blocking the formation of mRNA, and thus inhibiting the synthesis of DNA and RNA. In addition, epirubicin also has inhibitory effect on topoisomerase II. Compared with adriamycin, the effect of epirubicin is equal or slightly higher, but with less cardiotoxicity and myelotoxicity.

Although epirubicin has been widely used in chemotherapy regimen for the treatment of multiple types of solid cancer, due to lack of large-scale randomized clinical study, the use of epirubicin in the treatment of lymphoma is greatly limited and epirubicin has not been recommended in internationally recognized guidelines including NCCN, ESMO and ASH. There have been several studies using epirubicin for the treatment of lymphoma, which all indicated comparable efficacy and lower toxicity compared with adriamycin. Because CHOP regimen is often combined with targeted therapy, optimizing anthracyclines in CHOP regimen is quite important for reducing toxicity, especially replacing Adriamycin with epirubicin.

Up to present, there have been studies on elderly patients and low-risk young patients with DLBCL and the results have provided evidences to support R+CHOP21 as the first-line standard therapy for DLBCL. But there still lacks clinical studies on high-risk young DLBCL patients and the treatment for these kinds of patients often follows the therapy of above mentioned studies, and these lack strong support of evidenced medicine. Before the application of Rituximab, several studies have suggested that increasing dosage strength of anthracyclines may bring benefits in overall survival to patients. After the introduction of Rituximab in the treatment of DLBCL, although Rituximab significantly promote overall survival of low-risk patients, young high-risk patients have not been studied.

Based on above background and current knowledge gap, this clinical study shall focus on newly pathologically diagnosed young medium/high-risk Chinese DLBCL patients and investigate whether enhanced epirubicin dosage strength shall achieve higher complete remission rate and longer overall survival.

OBJECTIVES:

1. Evaluate and compare the efficacy of high-dose epirubicin (90mg/m2) and standard-dose epirubicin (75mg/m2) in R±CEOP chemotherapy regimen.
2. Assess toxicity profile of R±CEOP chemotherapy regimen at different dosage of epirubicin, especially difference in cardiotoxicity and hematological toxicity between R±CEOP90 and R±CEOP75.
3. Assess the influence of R±CEOP90 and R±CEOP75 on long-term survival of newly diagnosed young patients with medium/high-risk diffuse large B-cell lymphoma.

OUTLINE:

Included patients shall be randomly divided into 2 groups: high-dose epirubicin group (90mg/m2) and standard-dose epirubicin group (75mg/m2) given intravenously on Day 1 of each cycle for totally 6 cycles. Patients with CD20 positive proven by pathological examination in both groups shall receive Rituximab. Except for the difference in epirubicin dosage, the administration of Cyclophosphamide, Vincristine and Prednisolone shall follow standard chemotherapy regimen.

Screening shall be completed within 4 weeks before the administration of study drugs. For included patients, treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. During treatment of study drugs, the tests and procedures shall be performed within the first 3 days of each cycle: serum chemistry test, hematological test and body weight measurement. Physical examination, vital sign and WHO performance and ECOG score shall be performed or assess before the administration of study drugs on Day 1 of each cycle. At the end of Cycle 3, 6 and 8 (if applicable) (±14days), physical examination, CT or MRI or PET examination shall be performed. If necessary, bone marrow assessment shall also be performed.

End-of-treatment visit shall be conducted within 4-5 weeks after the last administration of study drug. Patients experiencing toxicity or side effects shall be assessed within 4 weeks after withdrawal of study drugs. After completion of study treatment, patients who have not shown signs of disease progression shall be followed up for 2 year until disease progression, start treatment for another disease or death. Follow-up visit shall be conducted every 12±2 weeks and tumor assessment shall be performed (including neck, chest, abdomen, and pelvis CT or MRI).

PROJECTED ACCRUAL: A total of 408 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. All newly diagnosed patients with histologically proven diffuse large B cell lymphoma (DLBCL);
2. There is at least one measurable tumor mass (physical examined long diameter of mass over 2 cm, or 5mmCT-scanned long diameter of mass over 1.5cm and short diameter over 1.0cm);
3. Male or female patients aged no younger than 18 and no elder than 60 years old;
4. aaIPI≥2 (LDH > normal +ECOG ≤2 + stage III-IV);
5. No involvement of the central nervous system;
6. ECOG score ≤ 2 points and expected survival ≥3 months;
7. During the study period, female subjects must be in menopause, or sterilization or willing to take contraceptive measures. Women with childbearing potential must use medically acceptable contraceptive method and agree to use this contraceptive method 2 weeks before treatment of the study drug, during study drug treatment and 3 months after the completion of study drug treatment;
8. Male subjects are required to take contraceptive measures and agree to use this contraceptive method 2 weeks before treatment of the study drug, during study drug treatment and 3 months after the completion of study drug treatment.
9. The subjects must be able to understand the study and are willing to participate in the study and sign informed consent;
10. The subjects must be able and willing to follow the research plan
11. Echocardiography measured LVEF ≥ 50%
12. Satisfied hematological function (based on the investigator's judgment, except for the DLBCL abnormal conditions) is defined as follows: Hemoglobin ≥9g/dl; absolute neutrophil count ≥1.5 * 10^9/L; platelet count ≥75 * 10^9/L

    -

Exclusion Criteria:

1. Primary central nervous system tumors or central nervous system metastasis;
2. previous drug induced cardiotoxicity > =CTCAE 3.0 Grade 2;
3. Complicated with serious heart disease which may affect this clinical study (e.g., heart failure [New York Heart Association NYHA Class III or IV, or left ventricular ejection fraction LVEF<50%] or with disease history of following diseases: QTc prolongation of clinical significance (for male patients, QTc over 450ms; for female patients, QTc over 470ms), ventricular tachycardia (VT) , atrial fibrillation (AF), heart block, myocardial infarction (MI) within 1 years, congestive heart failure (CHF) and coronary heart disease with symptoms requiring drug treatment;
4. Diagnosis of other malignancies other than diffuse large B cell lymphoma (DLBCL);
5. Mental disorders affecting compliance;
6. Unable to obtain informed consent;
7. Previously have received DLBCL treatment, except for biopsy or local radiotherapy;
8. Patients are pregnant or lactating women;
9. Patients have severe infections, medical conditions or psychiatric conditions, and investigators believe that this condition may interfere with the purpose of the study;
10. Patients with known positive human immunodeficiency virus (HIV), active hepatitis B, or active hepatitis C (positive for anti-HCV antibodies);
11. Existence of following laboratory abnormalities (unless any of these abnormalities are due to underlying lymphoma):

    1. Creatinine was greater than 1.5 folds of upper limit of normal (ULN) (except that creatinine clearance is within normal range) or calculated creatinine clearance<40 mL/min (using Cockcroft - Gault formula)
    2. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 folds of ULN
    3. Total bilirubin ≥1.5 folds of ULN: if total bilirubin ≤ 3 folds of ULN, patients with diagnosed Gilbert's disease can be included
12. In the absence of anticoagulant therapy, the international normalized ratio (INR) > 1.5 folds of ULN
13. In lupus patients without anticoagulant drug treatment, partial thromboplastin time (PTT) and activated partial thromboplastin time (aPTT) > 1.5 folds of ULN
14. Investigators decide that the patient is not suitable for this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 408 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 2 years
  Percentage of Complete remission (CR), Unconfirmed Complete Remission (CRu) and Partial remission (PR), referred to 2007 Cheson's Response Criteria for Lymphoma

SECONDARY OUTCOMES:
Time to response (TRR) | From date of drug administration until the date of the first remission (including Complete remission, Unconfirmed Complete Remission and Partial remission, whichever came first), assessed up to 2 years
  The time from drug administration to the first remission (including the first PR, CRu and CR)
Duration of response (DOR) | From date of the first remission until the date of first documented progression, assessed up to 2 years
  The time from remission to the first disease progression
Progression-free survival (PFS) | From date of drug administration until the date of progression disease or death, whichever came first, assessed up to 2 years
  The time from drug administration to the first progression disease or death
Overall survival(OS) | From date of drug administration until the date of death, assessed up to 2 years
  The time from drug administration to death

CONTACTS AND LOCATIONS:
Overall Officials: Jifeng Feng, M.D., Principal Investigator — Jiangsu Cancer Institute and Hospital
Locations (9):
- China (9):
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - Jiangyin People's hospital, Jiangyin, Jiangsu
  - Nanjing General Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Jiangsu Cancer Institute and Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - Wuxi People's hospital, Wuxi, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Economopoulos T, Dimopoulos MA, Mellou S, Pavlidis N, Samantas E, Nicolaides C, Tsatalas C, Papadopoulos A, Papageogriou E, Papasavvas P, Fountzilas G. Treatment of intermediate- and high-grade non-Hodgkin's lymphoma using CEOP versus CNOP. Eur J Haematol. 2002 Mar;68(3):135-43. doi: 10.1034/j.1600-0609.2002.01620.x. PMID 12068793
- [Background] Rossini F, Terruzzi E, Perego D, Miccolis I, Rivolta F, Manca E, Pogliani EM. Long-term follow-up of patients with intermediate or high-grade non-Hodgkin lymphoma treated with a combination of cyclophosphamide, epirubicin, vincristine, and prednisone. Cancer. 2004 Jan 15;100(2):350-5. doi: 10.1002/cncr.11907. PMID 14716771
- [Background] Chim CS, Kwong YL, Lie AK, Lee CK, Liang R. CEOP treatment results and validity of the International Prognostic Index in Chinese patients with aggressive non-Hodgkin's lymphoma. Hematol Oncol. 1998 Sep;16(3):117-23. doi: 10.1002/(sici)1099-1069(199809)16:33.0.co;2-0. PMID 10235070
- [Background] Lambertenghi Deliliers G, Butti C, Baldini L, Ceriani A, Lombardi F, Luoni M, Montalbetti L, Pavia G, Pinotti G, Pogliani E, et al. A cooperative study of epirubicin with cyclophosphamide, vincristine and prednisone (CEOP) in non-Hodgkin's lymphoma. Haematologica. 1995 Jul-Aug;80(4):318-24. PMID 7590500
- [Background] Coiffier B, Lepage E, Briere J, Herbrecht R, Tilly H, Bouabdallah R, Morel P, Van Den Neste E, Salles G, Gaulard P, Reyes F, Lederlin P, Gisselbrecht C. CHOP chemotherapy plus rituximab compared with CHOP alone in elderly patients with diffuse large-B-cell lymphoma. N Engl J Med. 2002 Jan 24;346(4):235-42. doi: 10.1056/NEJMoa011795. PMID 11807147
- [Background] Pfreundschuh M, Schubert J, Ziepert M, Schmits R, Mohren M, Lengfelder E, Reiser M, Nickenig C, Clemens M, Peter N, Bokemeyer C, Eimermacher H, Ho A, Hoffmann M, Mertelsmann R, Trumper L, Balleisen L, Liersch R, Metzner B, Hartmann F, Glass B, Poeschel V, Schmitz N, Ruebe C, Feller AC, Loeffler M; German High-Grade Non-Hodgkin Lymphoma Study Group (DSHNHL). Six versus eight cycles of bi-weekly CHOP-14 with or without rituximab in elderly patients with aggressive CD20+ B-cell lymphomas: a randomised controlled trial (RICOVER-60). Lancet Oncol. 2008 Feb;9(2):105-16. doi: 10.1016/S1470-2045(08)70002-0. Epub 2008 Jan 15. PMID 18226581
- [Background] Recher C, Coiffier B, Haioun C, Molina TJ, Ferme C, Casasnovas O, Thieblemont C, Bosly A, Laurent G, Morschhauser F, Ghesquieres H, Jardin F, Bologna S, Fruchart C, Corront B, Gabarre J, Bonnet C, Janvier M, Canioni D, Jais JP, Salles G, Tilly H; Groupe d'Etude des Lymphomes de l'Adulte. Intensified chemotherapy with ACVBP plus rituximab versus standard CHOP plus rituximab for the treatment of diffuse large B-cell lymphoma (LNH03-2B): an open-label randomised phase 3 trial. Lancet. 2011 Nov 26;378(9806):1858-67. doi: 10.1016/S0140-6736(11)61040-4. PMID 22118442
- [Background] Basaran M, Bavbek ES, Sakar B, Eralp Y, Alici S, Tas F, Yaman F, Dogan O O, Camlica H, Onat H. Treatment of aggressive non-Hodgkin's lymphoma with dose-intensified epirubicin in combination of cyclophosphamide, vincristine, and prednisone (CEOP-100): a phase II study. Am J Clin Oncol. 2001 Dec;24(6):570-5. doi: 10.1097/00000421-200112000-00008. PMID 11801756
- [Background] Pronzato P, Lionetto R, Botto F, Pensa F, Tognoni A. High-dose intensity cyclophosphamide, epidoxorubicin, vincristine and prednisone by shortened intervals and granulocyte colony-stimulating factor in non-Hodgkin's lymphoma: a phase II study. Br J Cancer. 1998 Sep;78(6):777-80. doi: 10.1038/bjc.1998.578. PMID 9743300
- [Background] Zinzani PL, Mazza P, Gherlinzoni F, Zanchini R, Bocchia M, Aitini E, Cavazzini G, Amurri B, Gobbi M, Tura S. CEOP regimen in the treatment of advanced low-grade non-Hodgkin's lymphomas: preliminary report. Tumori. 1990 Dec 31;76(6):533-6. doi: 10.1177/030089169007600603. PMID 2284688
- [Background] Abate G, Comella P, Di Pietro N, Ganzina F, Pergola M, Silvestro P, Basso A, Salvatore M, Zarrilli D. Epirubicin in combination chemotherapy in the treatment of advanced stage non-Hodgkin's lymphomas. Tumori. 1987 Feb 28;73(1):43-7. doi: 10.1177/030089168707300108. PMID 3469805